CLINICAL TRIAL: NCT04667078
Title: REperfusion With P2Y12 Inhibitors in Addition to mEchanical thRombectomy for perFUsion Imaging Selected Acute Stroke patiEnts (REPERFUSE)
Brief Title: REperfusion With P2Y12 Inhibitors in Addition to mEchanical thRombectomy for perFUsion Imaging Selected Acute Stroke patiEnts
Acronym: REPERFUSE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMI_2020_35
Record Dates: First submitted 2020-11-24; First posted 2020-12-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemia
MeSH Terms: interventions — cangrelor

STUDY DESIGN:
Intervention Model Description: experimental group will be treated by P2Y12 inhibitor (cangrelor) in addition to MT and BMM
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cangrelor group (Experimental): treated by P2Y12 inhibitor (cangrelor) in addition to MT and BMM. The dose of cangrelor will be started with a 30 micrograms/kg IV bolus over 1 minute right after randomization and before MT. The bolus will be immediately followed with 4 micrograms/kg/min IV infusion for the duration of MT up to 4 hours. Cangrelor infusion will be stopped at the end of the MT procedure and will not go further 4 hours. Transition to oral antiplatelet therapy will be possible 1 hour after cangrelor infusion discontinuation. No other anti-thrombotic drug is authorized during cangrelor infusion. MT technique choice is left to the investigator decision.
  Interventions: Drug: Cangrelor
- Best medical management group (Active Comparator): treated by BMM associated to MT. Anti-thrombotic including alteplase are authorized if they follow the recommendations of the international guidelines. If alteplase infusion is given, no other anti-thrombotic drug is allowed for the following 24 hours. MT technique choice is left to the choice of the investigator.
  Interventions: Other: best medical management

INTERVENTIONS:
Drug: Cangrelor — administration of cangrolor by iv befor thrombectomy
  Arms: Cangrelor group
Other: best medical management — used yhe best medical management
  Arms: Best medical management group

SUMMARY:
The main objective is to evaluate the efficacy of IV administration of the P2Y12 inhibitor (cangrelor) in addition to mecanich thrombectomy and WMD versus mecanich thrombectomy and WMD alone on the functional prognosis at 3 months, in patients with acute ischemic stroke eligible for mecanich thrombectomy on the basis of infusion imaging between 0 and 24 hours after the onset of symptoms.

DETAILED DESCRIPTION:
The emergent reperfusion of the ischemic penumbra is the goal of acute ischemic stroke (AIS) treatment. Mechanical thrombectomy (MT) may be proposed up to 6 hours and from 6 to 24 hours after stroke onset if multimodal imaging demonstrates the presence of a substantial ischemic penumbra.

Despite the major benefit associated with MT, more than half of patients will remain disabled at 3 months. The rate of complete reperfusion after MT appears to be a major factor affecting functional outcome. However, this rate of complete reperfusion is only achieved in 50 % of the patients due to, at least in part, distal microcirculatory impairment and or erratic emboli.

In coronary artery disease, new antiplatelet agents, with a very short half-life, such as P2Y12 inhibitors (P2Y12I), have been shown to reduce in-stent thrombosis, myocardial infarction and death. The IV route for P2Y12 inhibitors administration is adapted to the stroke population who has frequently dysphagia that prevents per os drug administration. In addition, the very short half-life of the drug is quite interesting for the management of hemorrhagic complications or emergent surgical interventions and early antithrombotic secondary prevention initiation.

Hypothesis: subgroup of patients treated from 0 to 24 hours after onset with a demonstrated ischemic penumbra on perfusion imaging, the administration of P2Y12I in addition to MT and best medical management (BMM) may increase reperfusion rates and improve functional outcome compared to MT with BMM alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Anterior circulation intracanial large artery occlusion isolated (Intracranial ICA and/or MCA) proved on CTA or MRA.
* Symptoms onset < 24h at imaging
* Indication for MT and fulfillment of the following brain imaging criteria :

  1. Perfusion imaging: An initial infarct volume (ischemic core on DWI or CTP calculated by the RAPID software) of less than 70 ml, a ratio between the critically hypoperfused lesion volume (calculated by RAPID with a TMax>6s) and initial infarct volume of 1.8 or more, and an absolute difference between those 2 volumes of 15 ml or more.

     OR (if perfusion imaging not available or uninterpretable) :
  2. CORE CLINICAL MISMATCH: Core calculated on DWI by RAPID, <25 mL if NIHSS 6-20 and <50 mL if NIHSS>20

     OR (if RAPID results are not considered reliable by the clinician) :
  3. CORE CLINICAL MISMATCH according to the clinician evaluation
* Pre-stroke mRS ≤ 2
* NIHSS ≥ 6

Exclusion Criteria:

* Contraindication to MT
* Patient over 80 years old with >10 microbleeds on pre-treatment MRI
* Pre-existing dependency with mRS ≥3.
* Known tandem ICA-MCA occlusions requiring stenting
* ASPECT<6 on NCCT or DWI-MRI
* Known hypersensitivity to cangrelor or to any of the excipients (mannitol, sorbitol)
* History of previous intracranial hemorrhage
* Evidence of active bleeding or acute trauma (fracture) on examination
* Recent surgery with a significant risk of bleeding
* VKA oral anticoagulation with INR >1.7
* Curative heparin or direct oral anticoagulants (DOACs) in previous 48 hours with specific DOAC dosage ≥50 ng/ml and abnormal thrombin time for patients on dabigatran or abnormal specific anti-Xa activity for patients on apixaban, edoxaban, or rivaroxaban
* Platelet count <100 000/ mm3
* Woman of childbearing age without a pregnancy test or with a positive serum pregnancy test
* Patient benefiting from a legal protection
* Non-membership of a national insurance scheme
* Opposition of the patient or (in case of inclusion as a matter of urgency) of the trustworthy person
* Participation in another study regarding AIS care interfering with this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Favorable functional evaluation at 3 month for patients with acute ischemic strocke treated by cangrelor. | 3 months
  The favorable functional outcome at 3 month will be evaluated using a modified Rankin Scale (mRS). The scale runs from 0 to 6, running from perfect health without symptoms to death (0: no symptoms, 3: Moderate disability. Requires some help, but able to walk unassisted, 6: Dead).

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU de Besançon, Besançon
  - Hôpital Pellegrin (CHU de Bordeaux), Bordeaux
  - Hospices civils de Lyon, Hôpital Pierre Wertheimer, Bron
  - Hôpital Salengro (CHU Lille), Lille
  - Hôpital Dupuytren (CHU Limoges), Limoges
  - CHU La Timone, Marseille
  - Hôpital Central (CHU de Nancy), Nancy
  - Hôpital Lariboisière AP-HP, Paris
  - Hôpital Pitié-Salpêtrière AP-HP, Paris
  - Hôpital Fondation A de Rothschild, Paris
  - CHU de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpital Purpan (CHU de Toulouse), Toulouse

IPD SHARING:
Plan to Share IPD: No